CLINICAL TRIAL: NCT07351500
Title: An Embedded Adaptive Randomized Controlled Trial of Corticosteroid Therapy for Severe Influenza Community-Acquired Pneumonia in Adults
Brief Title: Adaptive RCT of Corticosteroids for Severe Influenza Pneumonia in Adults
Acronym: CAPSTONE-IFV
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qingyuan Zhan (Other)
Responsible Party: Sponsor-Investigator, Qingyuan Zhan, Director, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-I2M-C&T-B-090C
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Influenza
Keywords: Influenza; community-acquired pneumonia; adaptive randomised controled trial; corticosteroids
MeSH Terms: conditions — Influenza, Human; Community-Acquired Pneumonia | interventions — Sodium Chloride; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (Placebo Comparator): Control group
  Interventions: Drug: Saline (0.9%, sterile, for infusion)
- Low dose steroids (Experimental): treated with low dose corticosteroids
  Interventions: Drug: low dose Methylprednisolone
- Moderate dose steroids (Experimental): treated with moderate dose corticosteroids
  Interventions: Drug: Moderate dose Methylprednisolone

INTERVENTIONS:
Drug: Saline (0.9%, sterile, for infusion) — Sailine as control
  Arms: Standard of Care
Drug: low dose Methylprednisolone — Methylprednisolone 0.5mg/kg ivgtt qd
  Arms: Low dose steroids
Drug: Moderate dose Methylprednisolone — Methylprednisolone 1.0mg/kg ivgtt qd
  Arms: Moderate dose steroids

SUMMARY:
Severe community-acquired pneumonia caused by influenza virus (hereafter referred to as severe influenza pneumonia) is a major etiology of community-acquired pneumonia leading to acute respiratory failure and ICU admission. It can rapidly progress to profound hypoxemia, acute respiratory distress syndrome (ARDS), and multiple organ dysfunction, and remains associated with substantial mortality. Although antiviral therapy-typically neuraminidase inhibitors-and well-established organ-support strategies are currently available, outcomes in a subset of critically ill patients remain poor despite antiviral and supportive care alone, with ICU mortality reported to be as high as 20-30%. Therefore, identifying effective adjunctive interventions beyond standard care to further reduce mortality in severe influenza pneumonia is of great clinical importance for improving outcomes in critically ill patients and alleviating the burden on families and society.

However, the use of systemic corticosteroids in influenza-associated community-acquired pneumonia (CAP) has long been highly controversial. Multiple studies have suggested that corticosteroid therapy may increase mortality among patients with H1N1 influenza. During the early phase of the COVID-19 pandemic, treatment strategies drew on this evidence and generally advised caution regarding corticosteroid use; subsequently, randomized controlled trials (RCTs) such as RECOVERY and REMAP-CAP demonstrated that low-dose corticosteroids (e.g., dexamethasone 6 mg/day) reduce mortality in patients with pneumonia requiring oxygen therapy. Recently, the U.S. Centers for Disease Control and Prevention (CDC) has emphasized the urgent need for RCTs evaluating low- to moderate-dose corticosteroids or other immunomodulatory agents to clarify their role in the management of influenza-associated CAP. Collectively, these observations underscore the urgency of pathogen-directed anti-inflammatory strategies for CAP-associated acute respiratory failure.

Accordingly, we plan to conduct an adaptive, randomized, open-label, controlled trial to evaluate the efficacy and safety of adjunctive corticosteroid regimens at different doses, in addition to early standard supportive care (including guideline-concordant antiviral therapy and organ support), for reducing mortality in patients with severe influenza pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Admission to the Intensive Care Unit (ICU).
* Meeting the diagnostic criteria for community-acquired pneumonia (CAP).
* Meeting at least one of the major diagnostic criteria for severe pneumonia:

  (i) Requirement for endotracheal intubation and mechanical ventilation;

(ii) Septic shock requiring vasopressor therapy after adequate fluid resuscitation.

-Or simultaneously fulfilling three of the minor criteria:

(i) Respiratory rate ≥ 30 breaths/min;

(ii) PaO₂/FiO₂ ≤ 250 mmHg;

(iii) Multilobar infiltrates;

(iv) Altered mental status and/or disorientation;

(v) Blood urea nitrogen ≥ 20 mg/dL (7.12 mmol/L);

(vi) Leukopenia (white blood cell count < 4 × 10⁹/L);

(vii) Thrombocytopenia (platelet count < 100 × 10⁹/L);

(viii) Hypothermia (core temperature < 36 °C);

(ix) Hypotension (systolic blood pressure < 90 mmHg) requiring aggressive fluid resuscitation.

* Confirmed influenza virus etiology: at least one positive nucleic acid test (RT-PCR/PCR) or next-generation sequencing (NGS) result for influenza virus in respiratory specimens (respiratory secretions, throat swabs, or bronchoalveolar lavage fluid).
* Severe community-acquired pneumonia (SCAP) patients admitted to the emergency department/ward/ICU due to respiratory failure within < 72 hours.
* Signed informed consent.

Exclusion Criteria:

* Patients receiving vasopressor therapy for septic shock at the time of enrollment.
* Terminally ill patients (expected survival <30 days, e.g., advanced malignancy).
* Clinical history suggesting overt aspiration.
* Documented active gastrointestinal bleeding.
* Presence of cystic fibrosis, obstructive pneumonia, active influenza, pulmonary tuberculosis, or fungal infection.
* Active viral hepatitis or active herpesvirus infection.
* Bone marrow suppression or HIV infection.
* Refusal of mechanical ventilation and endotracheal intubation.
* Uncontrolled hyperglycemia (diabetic ketoacidosis with blood ketones >3 mmol/L, or hyperosmolar hyperglycemic state with blood glucose >33.3 mmol/L and elevated osmolality).
* Known allergy to corticosteroids.
* Patients requiring anti-inflammatory corticosteroids or replacement hydrocortisone for any reason, or those already receiving prednisone >15 mg/day (or equivalent dose of another corticosteroid).
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
28-day all cause mortality | 28 days from inclusion

IPD SHARING:
Plan to Share IPD: Undecided